CLINICAL TRIAL: NCT05569343
Title: Risk Factors for Achieving Textbook Outcome After Laparoscopic Duodenum-preserving Total Pancreatic Head Resection: a Retrospective, Observational Study
Brief Title: Risk Factors for Achieving TO After LDPPHR-t
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor in Surgery, Chief Physician, Director of Surgical Supervision Department, Deputy Director of Institute of Hepatobiliary&Pancreatic, Director of Department of Biliary-Pancreatic Surgery, Tongji Hospital
Other Study IDs: TJDBPS12
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Neoplasm of Uncertain Behavior Head
Keywords: Textbook outcome; Risk factors; Endoscopic nasobiliary drainage; Total pancreatic head resection; Duodenum-preserving; Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Textbook outcome group: Achieving textbook outcome after laparoscopic duodenum-preserving total pancreatic head resection
  Interventions: Other: No intervention
- Non-Textbook outcome group: Not achieving textbook outcome after laparoscopic duodenum-preserving total pancreatic head resection
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any intervention

SUMMARY:
This is a single, retrospective, observational study to investigate the risk factors for achieving textbook outcome after laparoscopic duodenum-preserving total pancreatic head resection.

DETAILED DESCRIPTION:
Increasing numbers of benign or low-grade malignant neoplasms at the head of pancreas are being diagnosed due to computed tomography (CT), magnetic resonance imaging (MRI) and endoscopic ultrasonography (EUS). Laparoscopic duodenum-preserving total pancreatic head resection (LDPPHR-t) has been accepted as a valid alternative treatment for benign and low-grade malignant neoplasms at the head of the pancreas. The evaluation of quality of LDPPHR-t is important for surgeons to improve surgical quality. Currently, the evaluation of surgical quality mainly depends on some single outcome indicators, such as morbidity, mortality, readmission rate, or hospital stay. These single outcome indicators are difficult to accurately reflect the overall surgical quality and the composite outcome measures may be better than single outcome indicators. Textbook outcome (TO) is such a composite concept and is realized when all the requirements after operation are achieved according to the "all or none" principle. TO reflects the ideal surgical outcome and is a multidimensional measure for surgical quality assurance. However, the risk factors for achieving TO after LDPPHR-t is unknown and no relevant articles have been reported so far. The objective of study was to identify the risk factors for achieving TO after LDPPHR-t.

ELIGIBILITY:
Inclusion Criteria:

1. Patients underwent laparoscopic duodenum-preserving total pancreatic head resection.
2. Aged 18 to 75 years old.

Exclusion Criteria:

1. Peritoneal seeding or metastasis to distant sites.
2. Incomplete clinical data.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent laparoscopic duodenum-preserving total pancreatic head resection in the department of Biliary-Pancreatic Surgery of Tongji Hospital from May 2020 to December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
postoperative complications | up to 90 days
  The postoperative complications were graded into mild complications and severe complications according to the Clavien-Dindo classification of surgical complications, including postpancreatectomy hemorrhage, postoperative pancreatic fistula , and bile leakage.

SECONDARY OUTCOMES:
Operation time | Intraoperative
  Operation time defined as the time from skin incision or trocar placement to complete skin closure
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss recorded by the anesthetist using a vacuum system
Readmission | up to 30 days
  Readmission defined as any readmission within 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, MD, Study Director — Department of Biliary-Pancreatic Surgery, Affiliated Tongji Hospital
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China